CLINICAL TRIAL: NCT00591461
Title: A Prospective Study on the Interobserver Agreement of Endoscopic Barrett's Esophagus
Brief Title: Study of Endoscopic Barrett's Esophagus Diagnosis
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00003558
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Barrett's Esophagus; GERD
Keywords: Barrett's Esophagus; Upper Endoscopy; Esophageal biopsies; Accuracy; Interobserver Agreement
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Esophageal biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Study participants must be older than 18 years of age who are having an endoscopy performed to evaluate symptoms of GERD such as heartburn, acid taste in the mouth, dysphagia, dyspepsia, or those who are having a screening/surveillance exam for BE.

SUMMARY:
Barrett's esophagus (BE) is a condition that often occurs in patients who have had GERD for a long time. The researchers are interested in BE because it can sometimes become a cancer in the esophagus. The way that we currently diagnose BE is by performing an upper endoscopy and looking for a change in the color of the esophagus. This color change may represent BE. If the doctor sees this, he/she may take biopsies of this area.

Studies have shown that making the diagnosis of BE can be hard to make. One of the reasons why this may be is because doctors may interpret what they see differently during the procedure. In other words, they may see an esophagus that appears normal in color or abnormal in color.

The purpose of this study is to compare two doctors' impressions of the appearance of the esophagus during a single endoscopy procedure.

ELIGIBILITY:
Inclusion Criteria:

* History of (h/o) GERD
* Upper GI symptoms such as acid taste in mouth, dysphagia, dyspepsia
* Screening or surveillance exam for BE

Exclusion Criteria:

* Unable to consent
* History of esophageal varices

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants must be older than 18 years of age who are having an endoscopy performed to evaluate symptoms of GERD such as heartburn, acid taste in the mouth, dysphagia, dyspepsia, or those who are having a screening/surveillance exam for BE.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the interobserver variability in the presence of columnar epithelium as well as the measured lengths. | one endoscopy visit

SECONDARY OUTCOMES:
frequency of pathology-confirmed BE | one endoscopy visit
variables that predict endoscopic interobserver agreement and path-confirmation | one endoscopy visit

CONTACTS AND LOCATIONS:
Overall Officials: Glenn M Eisen, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - OHSU, Portland, Oregon
  - PVAMC, Portland, Oregon

REFERENCES:
- [Background] Eloubeidi MA, Provenzale D. Does this patient have Barrett's esophagus? The utility of predicting Barrett's esophagus at the index endoscopy. Am J Gastroenterol. 1999 Apr;94(4):937-43. doi: 10.1111/j.1572-0241.1999.990_m.x. PMID 10201460
- [Background] Padda S, Ramirez FC. Accuracy in the diagnosis of short-segment Barrett's esophagus: the role of endoscopic experience. Gastrointest Endosc. 2001 Nov;54(5):605-8. doi: 10.1067/mge.2001.118714. PMID 11677477
- [Background] Kim SL, Waring JP, Spechler SJ, Sampliner RE, Doos WG, Krol WF, Williford WO. Diagnostic inconsistencies in Barrett's esophagus. Department of Veterans Affairs Gastroesophageal Reflux Study Group. Gastroenterology. 1994 Oct;107(4):945-9. PMID 7926484
- [Background] Meining A, Ott R, Becker I, Hahn S, Muhlen J, Werner M, Hofler H, Classen M, Heldwein W, Rosch T. The Munich Barrett follow up study: suspicion of Barrett's oesophagus based on either endoscopy or histology only--what is the clinical significance? Gut. 2004 Oct;53(10):1402-7. doi: 10.1136/gut.2003.036822. PMID 15361485
- [Background] Guda NM, Partington S, Vakil N. Inter- and intra-observer variability in the measurement of length at endoscopy: Implications for the measurement of Barrett's esophagus. Gastrointest Endosc. 2004 May;59(6):655-8. doi: 10.1016/s0016-5107(04)00182-8. PMID 15114308